CLINICAL TRIAL: NCT07156461
Title: A Pivotal, Interventional, Prospective, Multi-centre Clinical Investigation of Hearing Outcomes With the Osia 3 Sound Processor Compared to the Osia 2 Sound Processor in Adult Osia Implant Recipients With Mixed Hearing Loss, Conductive Hearing Loss or Single-Sided Deafness
Brief Title: Hearing Outcomes With the Osia 3 Sound Processor Compared to the Osia 2 Sound Processor in Adult Osia Implant Recipients
Acronym: SONUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5861
Record Dates: First submitted 2025-08-26; First posted 2025-09-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Mixed; Hearing Loss, Conductive; Single-Sided Deafness; Bone Conduction
Keywords: Bone Conduction
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Conductive

STUDY DESIGN:
Intervention Model Description: The investigation uses a repeated-measures, cross-over design where study recipients will be randomized into one of two groups (1:1 ratio)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cochlear™ Osia® 2 Sound Processor (Active Comparator): Participants randomized to group 1 will first receive a study Osia 2 Sound Processor to use at home for 1-2 weeks, before returning to the clinic to complete various assessments. These participants will then switch to the Osia 3 Sound Processor and complete the same protocol.
  Interventions: Device: Cochlear™ Osia® System (Osia® 2); Device: Cochlear™ Osia® System (Osia® 3)
- Cochlear™ Osia® 3 Sound Processor (Experimental): Participants randomized to group 2 will first receive a Osia 3 Sound Processor to use at home for 1-2 weeks, before returning to the clinic to complete various assessments. These participants will then switch to the Osia 2 Sound Processor and complete the same protocol.
  Interventions: Device: Cochlear™ Osia® System (Osia® 2); Device: Cochlear™ Osia® System (Osia® 3)

INTERVENTIONS:
Device: Cochlear™ Osia® System (Osia® 2) — Consists of Osia 2 Sound Processor, Osia 2 Sound Processor Magnets, and Osia Fitting Software 2.
Device: Cochlear™ Osia® System (Osia® 3) — Consists of Osia 3 Sound Processor, Osia 3 Sound Processor Magnets, Osia 3 Charger, and Osia Fitting Software 3.

SUMMARY:
The goal of this interventional study is to evaluate the clinical performance and sound quality of the Osia 3 Sound Processor and to demonstrate its superiority compared with the Osia 2 Sound Processor in adults with mixed hearing loss, conductive hearing loss, or single-sided deafness.

The main questions this study aims to answer are:

* Do the findings confirm the clinical performance of the Osia 3 Sound Processor?
* Is the Osia 3 Sound Processor superior compared to the Osia 2 Sound Processor?

Participants will:

* Undergo speech performance testing in both quiet and noisy environments
* Provide ratings for a self-reported questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a Cochlear Osia Implant (OSI100, OSI200, OSI300)
* Conductive or mixed hearing loss in the implanted ear. Bone conduction thresholds up to 65 dB HL (up to 40 dB HL at 0.5 kHz, up to 55 dB HL at 1kHz and up to 65 dB HL at 2 and 4 kHz) or Single-Sided Deafness in the implanted ear. The pure tone average air conduction hearing thresholds of the hearing ear should be better than or equal to 20 dB HL (measured at 0.5, 1, 2 and, 3 kHz).
* Aged 18 years or older, at time of consent.
* Minimum experience of 1 month with the Osia 2 Sound Processor.
* Fluent speaker in the language used to assess speech perception performance.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Ongoing infection at or around the sound processor area.
* Bilaterally implanted with a Cochlear Osia Implant.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Mean difference in speech reception threshold in noise with the Osia 3 Sound Processor, 1-2 weeks after fitting compared to the unaided condition at baseline | At Baseline (Day 0), Visit 1 (7-14 days after Baseline), and Visit 2 (7-14 days after Visit 1)
  Speech perception in noise will be assessed using the Australian Speech Test in Noise (AuSTIN) at the Australian sites and the Bamford-Kowal-Bench Speech-In-Noise (BKB-SIN) test at the US site. The AuSTIN uses BKB-SIN like target sentences presented in noise and comprises of 80 lists of 20 sentences each. The BKB-SIN test contains 18 list pairs of sentences, each containing 3-4 key words, presented at 65 dB SPL with adaptive noise levels. Both tests aim to determine the signal-to-noise ratio (SNR) at which 50% of the key words are correctly repeated. For the unaided and aided measurements, speech performance in noise will be measured with speech and noise presented from a front speaker, positioned at 1 m from the subject.

SECONDARY OUTCOMES:
Mean difference in the word recognition score in quiet with the Osia 3 Sound Processor measured at 65 dB SPL, 1-2 weeks after fitting compared to the unaided condition at baseline | At Baseline (Day 0), Visit 1 (7-14 days after Baseline), and Visit 2 (7-14 days after Visit 1)
  Speech perception in quiet will be measured using the consonant-nucleus-consonant (CNC) monosyllabic words presented at 65 dB SPL from the front speaker. The CNC word test consists of 30 lists each with 50 words per list. The goal of the speech perception assessment in quiet is to obtain the percentage of correctly repeated words in a list, i.e., the word recognition score.
Mean difference in the four-frequency sound field threshold average (PTA4, mean of sound field thresholds at 0.5, 1, 2, and 4 kHz) with the Osia 3 Sound Processor, 1-2 weeks after fitting compared to the unaided condition at baseline | At Baseline (Day 0), Visit 1 (7-14 days after Baseline), and Visit 2 (7-14 days after Visit 1)
  Thresholds in sound field will be measured using warble tones presented from a front speaker positioned at 1 m from the subject following the modified Hughson-Westlake procedure. Frequencies to be tested are 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000, and 8000 Hz.
Mean difference in speech perception in noise with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor measured at a fixed signal-to-noise ratio (SNR) of 0 dB SNR, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Speech perception in noise with a fixed SNR will be measured using the AzBio sentence test, which consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. The sentences will be presented at a fixed level of 65 dB SPL at a fixed SNR of 0 dB SNR using the accompanying noise stimulus. Each word in the sentence counts towards the overall score (percent correct). Speech will be presented from the front, while noise will be presented from the rear.
Mean difference in speech perception in noise with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor measured at a fixed signal-to-noise ratio (SNR) of +5 dB SNR, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Speech perception in noise with a fixed SNR will be measured using the AzBio sentence test, which consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. The sentences will be presented at a fixed level of 65 dB SPL at a fixed SNR of +5 dB SNR using the accompanying noise stimulus. Each word in the sentence counts towards the overall score (percent correct). Speech will be presented from the front, while noise will be presented from the rear.
Mean difference in the Speech Spatial and Qualities of Hearing Scale (SSQ-12) global score with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  The SSQ-12 involves a self-reported hearing function and the impact of hearing treatment in daily life across a variety of listening situations. It includes 3 subcategories: Speech Hearing, Spatial Hearing, and Qualities of Hearing, with each question rated on a Likert scale from 0-10 (minimum - maximum hearing abilities).
Mean difference in the word recognition score in quiet with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor measured at 50 dB SPL, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Speech perception in quiet will be measured using the consonant-nucleus-consonant (CNC) monosyllabic words presented at 50 dB SPL from the front speaker. The CNC word test consists of 30 lists each with 50 words per list. The goal of the speech perception assessment in quiet is to obtain the percentage of correctly repeated words in a list, i.e., the word recognition score.
Mean difference in the word recognition score in quiet with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor measured at 65 dB SPL, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Speech perception in quiet will be measured using the consonant-nucleus-consonant (CNC) monosyllabic words presented at 65 dB SPL from the front speaker. The CNC word test consists of 30 lists each with 50 words per list. The goal of the speech perception assessment in quiet is to obtain the percentage of correctly repeated words in a list, i.e., the word recognition score.
Mean difference in speech reception threshold in noise with the Osia 3 Sound Processor compared with the Osia 2 Sound Processor, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Speech perception in noise will be assessed using the Australian Speech Test in Noise (AuSTIN) at the Australian sites and the Bamford-Kowal-Bench-Speech in Noise (BKB-SIN) test at the US site. The AuSTIN uses BKB-SIN like target sentences presented in noise and comprises of 80 lists of 20 sentences each. The BKB-SIN test contains 18 list pairs of sentences, each containing 3-4 key words, presented at 65 dB SPL with adaptive noise levels. Both tests aim to determine the signal-to-noise ratio (SNR) at which 50% of the key words are correctly repeated. For the unaided and aided measurements, speech performance in noise will be measured with speech and noise presented from a front speaker, positioned at 1 m from the subject.
Mean difference in the four-frequency sound field threshold average (PTA4, mean of sound field thresholds at 0.5, 1, 2, and 4 kHz) with the Osia 3 Sound Processor compared to the Osia 2 Sound Processor, 1-2 weeks after fitting | At Visit 1 (7-14 days after Baseline) and Visit 2 (7-14 days after Visit 1)
  Thresholds in sound field will be measured using warble tones presented from a front speaker positioned at 1 m from the subject following the modified Hughson-Westlake procedure. Frequencies to be tested are 250, 500, 750, 1000, 1500, 2000, 3000, 4000, 6000 and 8000 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: PRS Specialist, Study Director — Cochlear Ltd
Locations (3):
- Cochlear Americas, Denver Research and Technology Lab, Denver, Colorado, United States
- Australia (2):
  - Cochlear Macquarie, Macquarie University, Sydney, New South Wales
  - HEARnet Clinical Studies, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No